CLINICAL TRIAL: NCT04905043
Title: A Phase 1, Single-center, Open-label, Fixed-sequence, 2-period Study in Healthy Adult Subjects to Evaluate the Effect of Gastric pH on Acalabrutinib Pharmacokinetics
Brief Title: A Study to Evaluate the Effect of Gastric pH on Acalabrutinib Pharmacokinetics (PK) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-HV-113
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Acalabrutinib; ACP-196; Gastric pH; Healthy participants; Pharmacokinetics; PK; Safety
MeSH Terms: interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SmartPill® + Acalabrutinib (Experimental): Participants will receive 1 SmartPill® capsule followed immediately by a single oral dose of acalabrutinib 100 mg capsule on Day 1 (Period 1) and Day 4 (Period 2). There will be 72 hours of washout between acalabrutinib dosing of each period.
  Interventions: Drug: Acalabrutinib; Drug: SmartPill®

INTERVENTIONS:
Drug: Acalabrutinib — Participants will receive a single oral dose of acalabrutinib 100 mg capsule on Day 1 (Period 1) and Day 4 (Period 2).
  Other Names: ACP-196
Drug: SmartPill® — Participnats will receive a single oral dose of wireless motility/pH capsule (SmartPill®) on Day 1 (Period 1) and Day 4 (Period 2).

SUMMARY:
This study will evaluate the effect of gastric pH on acalabrutinib pharmacokinetics in healthy participants.

DETAILED DESCRIPTION:
This is a 2-period study done under fasting conditions. Participants will receive an oral wireless motility/pH capsule (SmartPill®) followed immediately by a single 100 mg oral dose of acalabrutinib on Day 1 of Period 1 and Period 2 (ie, Day 1 and Day 4, respectively). There will be 72 hours of washout between Day 1 dosing of each period. Participants will be contacted approximately 14 days after the last dose of study drug for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Continuous nonsmoker who has not used nicotine-containing products for >= 3 months before the first dose.
* Body mass index (BMI) >= 18.0 and <= 32.0 kg/m^2 at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or ECGs, as deemed by the principal investigator. Liver function tests, and serum bilirubin, must be <= upper limit of normal range (ULN) at screening.
* Minimum of 1 bowel movement per day for >= 3 months before enrollment.
* Women must be of non-childbearing status and must have negative serum pregnancy test results.
* Men of reproductive potential to follow protocol defined contraception methods.

Exclusion Criteria:

* Participant is mentally or legally incapacitated, or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* Participant has any of the following contraindications for the SmartPill: A history of gastric bezoars, swallowing disorder, suspected or known strictures, fistulas or physiological/mechanical gastrointestinal (GI) obstruction, history of GI surgery within 3 months of administration, severe dysphagia to food or pills, Crohn's disease or diverticulitis, cardiac pacemakers or other implanted electromedical devices.
* History or presence of alcoholism or drug abuse within the past 2 years before screening
* History of bleeding diathesis
* History of gastric motility disorder for example delayed gastric emptying, dumping syndrome, or irritable bowel disease.
* History of constipation within the last year before enrollment
* Currently experiencing, or experienced within 2 weeks of enrollment, Grade 2 diarrhea
* Women who are pregnant or breastfeeding
* Positive urine drug or alcohol results at screening or check-in
* Positive urine cotinine at screening.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Seated blood pressure is < 90/40 mmHg or > 140/90 mmHg at screening.
* Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
* Have been on a diet incompatible with the on study diet, in the opinion of the principal investigator (PI), within the 28 days before the first dose of study drug, and throughout the study.
* Unable to refrain from or anticipates the use of protocol defined medications.
* History or presence of liver disease and clostridium difficile-associated diarrhea.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-03 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Effect of Gastric pH and Emptying Rate on Acalabrutinib PK Parameters (Area Under Concentration-time Curve [AUC] From Time 0 to Last Measurable Concentration, AUC From Time 0 to Infinity, Maximum Observed Plasma Concentration [Cmax], Time to Reach Cmax) | 0, 3, 8, and 17 minutes post-ingestion event time (IET) in Periods 1 and 2
Area Under the Plasma Concentration-time Curve From Time 0 to Time of Last Measurable Concentration (AUC0-last) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Maximum Observed Plasma Concentration (Cmax) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2

SECONDARY OUTCOMES:
Percent of AUC0-inf Extrapolated (AUC%extrap) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours (AUC0-6h) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Area Under the Plasma Concentration-time Curve From Time 0 to 12 Hours (AUC0-12h) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Time to Reach Maximum Observed Plasma Concentration (Tmax) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Apparent Terminal Elimination Rate Constant (λz) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Apparent Terminal Elimination Half-life (T1/2) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Apparent Total Plasma Clearance (CL/F) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Apparent Volume of Distribution (Vz/F) of Acalabrutinib | pre-dose; and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose in Periods 1 and 2
Incidences of Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) | Day 1 through 14 days after the last dose (approximately 1 month)
Incidences of Abnormal Vital Signs and Physical Examinations Reported as TEAEs | Day 1 to Day 5 for each participant
Incidences of Abnormal Electrocardiograms (ECGs) Reported as TEAEs | Day 1 to Day 5 for each participant
Incidences of Abnormal Clinical Laboratory Parameters Reported as TEAEs | Day 1 to Day 5 for each participant

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home